CLINICAL TRIAL: NCT05698186
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase III Efficacy and Safety Study of Thero2-01S22 add-on Therapy on Top of First-line Anti-HER2 Targeted Treatment of Patients With Metastatic Breast Cancer
Brief Title: Thero2-01S22 in HER2-positive Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-009
Record Dates: First submitted 2022-11-30; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: HER2-positive Breast Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1: Anti-HER2 targeted therapy containing regimen + Thero2-01S22 (Experimental): Patients will receive Thero2-01S22 at the recommended dose and induction therapy according to local practice with a taxane (docetaxel, paclitaxel, or nab-paclitaxel) or vinorelbine for 4 to 6 cycles in combination with pertuzumab and trastuzumab
  Interventions: Drug: Thero2-01S22
- Part 1: Anti-HER2 targeted therapy containing regimen + Placebo (Placebo Comparator): Patients will receive placebo and induction therapy according to local practice with a taxane (docetaxel, paclitaxel, or nab-paclitaxel) or vinorelbine for 4 to 6 cycles in combination with pertuzumab and trastuzumab
  Interventions: Drug: Placebo
- Part 2: Anti-HER2 targeted therapy containing regimen + Thero2-01S22 (Experimental): Patients will receive Thero2-01S22 at the confirmed dose and induction therapy according to local practice with a taxane (docetaxel, paclitaxel, or nab-paclitaxel) or vinorelbine for 4 to 6 cycles in combination with pertuzumab and trastuzumab
  Interventions: Drug: Thero2-01S22
- Part 2: Anti-HER2 targeted therapy containing regimen + Placebo (Placebo Comparator): Patients will receive placebo and induction therapy according to local practice with a taxane (docetaxel, paclitaxel, or nab-paclitaxel) or vinorelbine for 4 to 6 cycles in combination with pertuzumab and trastuzumab
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thero2-01S22 — Blinded recommended dose BID for three (3) consecutive days starting the day before anti-HER2 targeted therapy containing regimen, at cycle 1 and cycle 2
  Arms: Part 1: Anti-HER2 targeted therapy containing regimen + Thero2-01S22
Drug: Placebo — Blinded placebo BID for three (3) consecutive days starting the day before anti-HER2 targeted therapy containing regimen, at cycle 1 and cycle 2
  Arms: Part 1: Anti-HER2 targeted therapy containing regimen + Placebo
Drug: Thero2-01S22 — Blinded confirmed dose BID for three (3) consecutive days starting the day before anti-HER2 targeted therapy containing regimen, at cycle 1 and cycle 2
  Arms: Part 2: Anti-HER2 targeted therapy containing regimen + Thero2-01S22
Drug: Placebo — Blinded placebo BID for three (3) consecutive days starting the day before anti-HER2 targeted therapy containing regimen, at cycle 1 and cycle 2
  Arms: Part 2: Anti-HER2 targeted therapy containing regimen + Placebo

SUMMARY:
Trastuzumab and pertuzumab based regimen are the standard of care for patients with human epidermal growth factor receptor 2 (HER2) -positive metastatic breast cancer (MBC), significantly improving survival outcomes. However, an unmet medical need remain for patients with disease refractoriness and recurrence. Interestingly, HER2 over-expression is associated with upregulation of vascular endothelial growth factor (VEGF) in cancer cells in vitro and in vivo. Preclinical studies indicated that VEGF expression is positively regulated by HER2 signaling. In the clinical setting, HER2 over-expression correlated significantly with VEGF over- expression in samples from patients with breast cancer. There is, therefore, a biologic rationale for targeting both HER2 and VEGF pathways in patients with HER2-positive breast cancer.

PURPOSE: The hypothesis that justifies this research is that the addition of Thero2-01S22 as add-on therapy on top of first line anti-HER2 targeted treatment will improve the efficacy of anti-HER2 targeted containing regimen at the metastatic setting for breast cancer.

DETAILED DESCRIPTION:
This study is a two-part, multicenter, randomized, double-blind, placebo-controlled, Phase III trial.

Part 1 will confirm the recommended Phase III dose of Thero2-01S22 when administered as add-on therapy on top of first line anti-HER2 targeted treatment of patients with metastatic breast, with the aim to obtain about 15 evaluable participants in Thero2-01S22 group and 15 in the placebo group.

Part 2 will assess the efficacy of Thero2-01S22 treatment at the recommended dose when administered as add-on therapy on top of first line anti-HER2 targeted treatment of patients with metastatic breast. Approximately 290 participants will be randomized to receive Thero2-01S22 or Thero2-01S22 matching-placebo in combination with trastuzumab and pertuzumab.

Participants in both Part 1 and Part 2 will receive induction therapy according to local practice with a taxane (docetaxel, paclitaxel, or nab-paclitaxel) or vinorelbine for 4 to 6 cycles in combination with pertuzumab and trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged > 18
2. Metastatic setting of an histologically confirmed adenocarcinoma of the breast
3. Performance status = 0, 1 or 2
4. Metastatic disease requiring the initiation of an anti HER2 containing regimen
5. First line treatment for metastatic disease
6. Standard treatment including Trastuzumab and Pertuzumab in first line
7. Patients for whom a 3-month life expectancy is anticipated
8. Baseline LVEF value > 50%, measured cardiac MRI or by echocardiography (Simpson's method) or MUGA scan within 12 weeks before initiation of the treatment. According to HERCEPTIN SPCs.
9. Overexpression of HER2 in the invasive component of the primary tumor (3+ by ICH or 2+ with confirmation of positivity by FISH or CISH)
10. Informed consent form signed

Exclusion Criteria:

1. Patients not eligible for anti-HER2 therapy
2. Patients previously treated at the metastatic setting by systemic treatment
3. Serious cardiac illness or medical conditions disallowing administration of anti-HER2 therapy. According to HERCEPTIN and PERJETA SPCs.
4. Known hypersensitivity to trastuzumab, pertuzumab, Thero2-01S22, murine proteins or to any of the excipients.
5. Uncontrolled central nervous system metastatic lesion
6. Patients who, for social, geographic or psychological reasons, cannot be adequately followed up and/or are incapable of undergoing regular controls
7. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 320 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Part 1: confirm the recommended dose of Thero2-01S22 as add-on therapy on top of first line anti-HER2 targeted treatment of patients with metastatic breast for Part 2 | Week 6
  Incidence of adverse events considered possibly related to Thero2-01S22 that occur any time from the first dose intake of IMP or placebo to week 6.
Part 2: compare the effects of anti-HER2 targeted containing regimen with and without Thero2-01S22 in terms of Objective response rate (ORR) at week 6 | Week 6
  Objective response rate (ORR): Percentage of patients whose disease decreased (Partial Response, PR) and / or disappears (Complete Response, CR) after treatment, according to RECIST V1.1 criteria, Eisenhauer et al. 2009.

SECONDARY OUTCOMES:
Part 1: determine the safety of the recommended dose of Thero2-01S22as add-on therapy on top of first line anti-HER2 targeted treatment of patients with metastatic breast cancer | Week 6
  Safety: Incidence of adverse events per Common Terminology Criteria for Adverse Events (graded according to CTCAE) version 5.0 criteria from randomization to week 6
Part 1: determine the tolerability of the recommended dose of Thero2-01S22 as add-on therapy on top of first line anti-HER2 targeted treatment of patients with metastatic breast cancer in terms of dose interruption | Week 6
  Number of dose interruptions of Thero2-01S22 trastuzumab, pertuzumab, and induction chemotherapy. Assessment period: from randomization to week 6
Part 1: determine the tolerability of the recommended dose of Thero2-01S22 as add-on therapy on top of first line anti-HER2 targeted treatment of patients with metastatic breast cancer in terms of palatability | Week 6
  Palatability of oral Thero2-01S22 measured with visual analog scale. Assessment period: from randomization to week 6
Part 1: determine the tolerability of the recommended dose of Thero2-01S22 as add-on therapy on top of first line anti-HER2 targeted treatment of patients with metastatic breast cancer in terms of treatment duration | From randomization to Week 6
  Treatment duration (number of days) of therapy including Thero2-01S22 trastuzumab, pertuzumab, and induction chemotherapy. Assessment period: from randomization to week 6
Part 1: characterize exposure of Thero2-01S22 when administered as add-on therapy on top of first line anti-HER2 targeted treatment of patients with metastatic breast | PK samples at day 1 of cycle 1 and cycle 2(each cycle is 21 days): before IMP or placebo intake, and at 5, 10, 15, 60, 120, 160 minutes after the intake
  Determination of Area Under Curve (AUC) after oral Thero2-01S22 administration. PK samples to be collected at day 1 of cycle 1 and cycle 2 (each cycle is 21 days): before IMP or placebo intake, and at 5, 10, 15, 60, 120, 160 minutes after the intake
Part 1: characterize exposure of Thero2-01S22 when administered as add-on therapy on top of first line anti-HER2 targeted treatment of patients with metastatic breast | PK samples at day 1 of cycle 1 and cycle 2(each cycle is 21 days): before IMP or placebo intake, and at 5, 10, 15, 60, 120, 160 minutes after the intake
  Determination of Maximum Plasma Concentration (Cmax) after oral Thero2-01S22 administration. PK samples to be collected at day 1 of cycle 1 and cycle 2 (each cycle is 21 days): before IMP or placebo intake, and at 5, 10, 15, 60, 120, 160 minutes after the intake
Part 1: evaluate preliminary efficacy of Thero2-01S22 when administered as add-on therapy on top of first line anti-HER2 targeted treatment of patients with metastatic breast cancer | Week 6
  Objective response rate (ORR): Percentage of patients whose disease decreased (Partial Response, PR) and / or disappears (Complete Response, CR) after treatment, according to RECIST V1.1 criteria, Eisenhauer et al. 2009.
  Calculated at week 6 after the last intake of IMP or placebo
Part 2: compare the effects of anti-HER2 targeted containing regimen with and without Thero2-01S22 in terms of Progression-Free Survival (PFS) | Up to 24 months
  Progression-Free Survival (PFS): defined as the time interval from the date of randomization to the date of progression.
  Events considered as progression include local or distant progression, appearance of a second cancer or death (all causes) whichever occurs first
Part 2: compare the effects of anti-HER2 targeted containing regimen with and without Thero2-01S22 in terms of Overall Survival (OS) | Up to 24 months
  Overall Survival (OS): defined as the time interval from the date of randomization to the date of death, regardless of disease progression
Part 2: compare the effects of anti-HER2 targeted containing regimen with and without Thero2-01S22 in terms of safety | Week 6 and up to the end of the study (24 months)
  Compare the effects of anti-HER2 targeted containing regimen with and without Safety: Incidence of treatment-related adverse events (AEs) and serious adverse events (SAEs) classified according to the CTCAE v5.0 criteria
Part 2: compare the effects of anti-HER2 targeted containing regimen with and without Thero2-01S22 in terms of cardiotoxicity in terms of decrease of Left Ventricular Ejection Fraction (LVEF) | From week 6 up to 24 months
  Decrease in Left Ventricular Ejection Fraction (LVEF) value compared to baseline according to the modality performed (ECG, MUGA, MRI)
Part 2: compare the effects of anti-HER2 targeted containing regimen with and without Thero2-01S22 in terms of cardiotoxicity in terms of cardiac toxicities revealed at physical examination | From week 6 up to 24 months
  Cardiac toxicities revealed at physical examination, graded according to CTCAE v5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Xavier PIVOT, MD, PhD, Study Chair — Institut de cancérologie Strasbourg Europe